CLINICAL TRIAL: NCT01398020
Title: Oral 2L Bi-PegLyte Versus 4L PegLyte Regimen for Outpatient Colonic Preparation: A Randomized, Non-Inferiority Open Trial
Brief Title: Comparing 2L Bi-Pegyte to 4L PegLyte Regiments for Outpatient Colonic Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H11-00688
Record Dates: First submitted 2011-07-14; First posted 2011-07-20 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Efficacy of Bowel Preparation; Ease of Bowel Preparation and Patient Tolerability
Keywords: Bowel Preparation; Patient comfort; Bi-Peglyte

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Standard bowel prep (Active Comparator): Subject will receive standard bowel prep prior to colonoscopy.
  Interventions: Drug: Standard Bowel Prep
- 2L Bi-Peglyte (Experimental): Subjects will be asked to take 2L Bi-Peglyte + 15mg bisacodyl for bowel prep the day before colonoscopy.
  Interventions: Drug: 2L Bi-Peglyte Bowel Prep

INTERVENTIONS:
Drug: Standard Bowel Prep — Subjects will be asked to take 4L of Peglyte the day prior to procedure.
  Arms: Standard bowel prep
Drug: 2L Bi-Peglyte Bowel Prep — Subjects will be asked to take 2L Bi-Peglyte and 15mg bisacodyl the day prior to procedure.
  Arms: 2L Bi-Peglyte

SUMMARY:
The investigators wish to compare the efficacy and patient tolerability of a preparation consisting of 2L Bi-Peglyte plus 15mg of bisacodyl vs the standard preparation of 4L Peglyte. The investigators hypothesize that 2L Bi-Peglyte with 15mg bisacodyl will show higher efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older
* Outpatient colonoscopy

Exclusion Criteria:

* constipation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference in Boston Bowel Preparation Scale between the two groups | 30 minutes
  This is an established rating scale to evaluate the quality of bowel prep. The ratings will be compared between the two groups.

SECONDARY OUTCOMES:
Difference in the number of participants who develop distress symptoms from bowel prep (and the type) between the two groups | 20 hours
  Number of participants who develop distress symptoms from bowel prep, and the type of distress symptoms will be compared between the two groups
Difference in the absolute number/percentage of participants in the two groups who find the bowel prep experience easy, acceptable, difficult, very difficult, or unable to complete. | 20
  Participants will be asked to rate their bowel prep experience (based on ease of use) on a Likert scale. The number of participants in each level will subsequently be quantified (n, %) and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Enns, MD, Principal Investigator — The University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada